CLINICAL TRIAL: NCT05387278
Title: Safety and Effectiveness of Placental Derived Exosomes and Umbilical Cord Mesenchymal Stem Cells in Moderate to Severe Acute Respiratory Distress Syndrome (ARDS) Associated With the Novel Corona Virus Infection (COVID-19)
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor request
Sponsor: Vitti Labs, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EW-01
Record Dates: First submitted 2022-05-16; First posted 2022-05-24 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: COVID-19 Acute Respiratory Distress Syndrome; Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Experimental/treatment arm (Experimental)
  Interventions: Drug: EV-Pure™ and WJ-Pure™
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: EV-Pure™ and WJ-Pure™ — The treatment consists of administration of WJ-Pure™ and EV-Pure™ plus standard care
  Arms: Experimental/treatment arm
Drug: Placebo — Cryopreservation media plus standard care
  Arms: Placebo

SUMMARY:
Recent advances have been made in prevention of the viral infection via vaccines but there is still need for effective treatment options for patients. Novel therapies need to be developed to further improve clinical outcomes. The biggest medical challenge in the response to COVID-19 is ARDS requiring hospitalization in an intensive care setting and ventilator dependence. Intravenously administered umbilical cord derived exosomes and stem cells have been reported in literature to alleviate pulmonary distress in such patients.

The purpose of this study is to explore the safety and benefits of intravenous administration of WJPure and EVPure in the treatment of COVID-19 patients with moderate to severe ARDS. .

DETAILED DESCRIPTION:
One of the hallmark features of the progression of COVID-19 is lung injury from the viral infection leading to potentially acute respiratory distress syndrome (ARDS) and respiratory failure requiring ventilator support. In patients who survive ARDS, regardless of the pathology, there is evidence that their long-term quality of life is adversely affected.

The rationale for the dose and dosing regimen proposed in this study is based on the safe administration and benefits of this treatment regimen reported to us last year by physicians trying to treat moderate to severe COVID-19 patients. In those reports, the intravenous route of administration was used. It has been reported that dosing every 2 days amplified the benefit of the combination of exosomes and mesenchymal stem cells. It has been suggested based on clinical experience that the exosomes and MSCs are complementary to one another as well as enhancing the innate abilities of both.

During the early days of the pandemic, intravenous infusion of a mixture of EV-Pure™ and WJ-Pure™ was reported to benefit hospitalized patients with moderate to severe COVID-19 related ARDS. This study is designed to systematically explore the risk and benefits of intravenous infusion of EV-Pure™ and WJ-Pure™ in the treatment of hospitalized COVID-19 patients with moderate to severe ARDS.

This is a proof of concept, double-blind, placebo-controlled trial to evaluate the safety and efficacy of intravenous infusion of EV-Pure™ and WJ-Pure™, versus placebo, for use in the treatment of moderate to severe ARDS related to COVID-19. This is an add-on treatment study; subjects will be allowed to take standard of care treatments available.

The study will have two arms (n=10 each):

1. Experimental/treatment arm: EV-Pure™ and WJ-Pure™ plus standard care
2. Placebo: Cryopreservation media plus standard care

The study duration would be 5 days of treatment plus 12 weeks follow up.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be eligible for enrollment in the study only if they meet the following criteria:

  1. Male or female, aged at 18 years (including) to 75 years old.
  2. Patient with a confirmed SARS-CoV-2 infection (by positive reverse-transcription polymerase chain reaction (RT-PCR) from nasopharyngeal sample or any other sample)
  3. Hospitalized with moderate to severe ARDS.
  4. Have ARDS or acute lung injury, comply with any of the following:

     i. Respiratory distress, Respiratory rate (RR) ≥ 30 times/min ii. Pulse oxygen saturation (SpO2) at rest ≤ 93% iii. Partial pressure of oxygen/fraction of inspired oxygen (PaO2/FiO2) ≤ 300mmHg
  5. If childbearing age: agree to practice effective birth control from screening until 12 weeks after the last study treatment.

Exclusion Criteria:

* Subjects will be ineligible for enrollment in the study if they meet any of the following criteria:

  1. Patient under invasive mechanical ventilation for more than 48 hours
  2. Allergic or hypersensitive to any of the ingredients.
  3. Pneumonia caused by bacteria, mycoplasma, chlamydia, legionella, fungi or other viruses.
  4. Obstructive HABP/VABP induced by lung cancer or other known causes.
  5. Carcinoid syndrome.
  6. History of long-term use of immunosuppressive agents.
  7. History of Class III or IV pulmonary arterial hypertension.
  8. Patient with chronic respiratory disease under oxygen therapy.
  9. Undergoing hemodialysis or peritoneal dialysis.
  10. Estimated or actual rate of creatinine clearance < 15 mL/min.
  11. History of moderate and severe liver disease (Child-Pugh score >12).
  12. History of deep venous thrombosis or pulmonary embolism within the last 3 years.
  13. Undergoing extracorporeal membrane oxygenation (ECMO) or high-frequency oscillatory ventilation support.
  14. Patient included in another ongoing interventional therapeutic trial.
  15. Pregnant or Lactating.
  16. Any condition of unsuitable for the study determined by Principal Investigator (PI).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-03-20 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
To Assess the safety of EV-Pure™ and WJ-Pure™ administration in patients exhibiting moderate to severe ARDS associated with COVID-19, compared to placebo. | 3 months
  Evaluate incidences of Treatment-Emergent Adverse Events following EV-Pure™ and WJ-Pure™ administeration in patients exhibiting moderate to severe ARDS associated with COVID-19 compared to placebo. Presence of adverse events in less than 10% of the study population, as a measure of safety
To assess the efficacy of EV-Pure™ and WJ-Pure™ compared to placebo, in patients with moderate to severe ARDS assoociated with COVID-19 | 3 Months
  Clinical data will be evaluated to determine if there were any significant changes in the COVID-19 symptoms in patients in the treated versus placebo groups. The following information will be collected to evaluate the effectiveness of the treatment at 4 weeks post- treatment:
  1. Discharged home on no supplemental oxygen
  2. Discharged home on supplemental oxygen
  3. Continued hospitalization on no oxygen
  4. Continued hospitalization on oxygen but not in ICU
  5. Continued hospitalization on oxygen in ICU (invasive and noninvasive ventilatory support)
  6. Death

SECONDARY OUTCOMES:
Time to clinical improvement | 3 months
  The following information will be collected from the subjects during the follow-up visits or calls:
  1. Medical history review
  2. Physical exam and vital signs
  3. Assessment for delayed adverse reactions
Overall Survival | 3 months
  Survival of the subjects in the 2 arms of the study
COVID-19 polymerase chain reaction (PCR) test result as negative | 3 months
  COVID-19 polymerase chain reaction (PCR) test result as negative in the subjects in the 2 arms of the study

CONTACTS AND LOCATIONS:
Locations (1):
- Kit Bartalos, Liberty, Missouri, United States